CLINICAL TRIAL: NCT01098474
Title: Safety and Immunogenicity Study of GSK Biologicals' Candidate Tuberculosis Vaccine (692342) When Administered to Healthy Infants
Brief Title: Safety and Immunogenicity Study of a Candidate Tuberculosis Vaccine in Healthy Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Aeras (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112899; 2012-004380-44 (EudraCT Number)
Record Dates: First submitted 2010-03-18; First posted 2010-04-02 (Estimated); Results first posted 2018-11-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Tuberculosis
Keywords: Tuberculosis vaccine
MeSH Terms: conditions — Tuberculosis | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SB692342 2 dose Group (Experimental): Subjects received two doses of SB692342 vaccine (0,5 mL), administered intramuscularly in the anterolateral region of the right thigh, 1 month apart, on a 0, 1 month schedule after having completed their primary EPI regimen.
  Interventions: Biological: GSK's investigational vaccine 692342
- SB692342 1 dose Group (Experimental): Subjects received one dose of SB692342 vaccine (0,5 mL), administered intramuscularly in the anterolateral region of the right thigh, at Month 0, after having completed their primary EPI regimen.
  Interventions: Biological: GSK's investigational vaccine 692342
- Control Menjugate Group (Active Comparator): Subjects received three doses of the control Menjugate™ vaccine (0,5 mL), administered intramuscularly in the anterolateral region of the right thigh, on a 0, 1, 7 months schedule. The first two doses were administered 1 month apart during the primary vaccination phase and the third dose was administered 6 months after the last primary vaccination dose.
  Interventions: Biological: Menjugate™
- SB692392 2 dose + Tritanrix + Prevnar + Polio Sabin Group (Experimental): Subjects received two doses of SB692342 vaccine (0,5 mL), administered intramuscularly in the anterolateral region of the right thigh, 1 month apart, concomintantly with the last two doses of the primary EPI regimen containing Tritanrix™ HepB+Hiberix™ vaccine, administered intramuscularly in the anterolateral region of the left thigh, Polio Sabin™ vaccine, administered orally, and Prevnar® vaccine, administered instramuscularly in the right arm, on a 0, 1, 2 months schedule.
  All subjects received a booster dose of the Tritanrix™ HepB+Hiberix™, Polio Sabin™ and Prevnar® vaccines approximately 1 year after their last dose.
  Interventions: Biological: GSK's investigational vaccine 692342; Biological: Tritanrix™ HB+Hib; Biological: Prevnar™; Biological: Polio Sabin™
- SB692392 1 dose + Tritanrix + Prevnar + Polio Sabin Group (Experimental): Subjects received one dose of SB692342 vaccine (0,5 mL), administered intramuscularly in the anterolateral region of the right thigh, concomitantly with the last dose of the primary EPI regimen containing Tritanrix™ HepB+Hiberix™ vaccine, administered intramuscularly in the anterolateral region of the left thigh, Polio Sabin™ vaccine, administered orally, and Prevnar® vaccine, administered intramuscularly in the right arm, on a 0, 1, 2 months schedule. All subjects received a booster dose of the Tritanrix™ HepB+Hiberix™, Polio Sabin™ and Prevnar® vaccines approximately 1 year after their last dose.
  Interventions: Biological: GSK's investigational vaccine 692342; Biological: Tritanrix™ HB+Hib; Biological: Prevnar™; Biological: Polio Sabin™
- Control Tritanrix + Prevnar + Polio Sabin Group (Active Comparator): Subjects received three doses of the primary EPI regimen containing Tritanrix™ HepB+Hiberix™ vaccine, administered in the anterolateral region of the left thigh, Polio Sabin™ vaccine, administered orally, and Prevnar® vaccine administered intramuscularly in the right arm, on a 0, 1, 2 months schedule. All subjects received a booster dose of the Tritanrix™ HepB+Hiberix™, Polio Sabin™ and Prevnar® vaccines approximately 1 year after their last dose.
  Interventions: Biological: Tritanrix™ HB+Hib; Biological: Prevnar™; Biological: Polio Sabin™

INTERVENTIONS:
Biological: GSK's investigational vaccine 692342 — Intramuscular, 1 or 2 doses
  Arms: SB692342 1 dose Group; SB692342 2 dose Group; SB692392 1 dose + Tritanrix + Prevnar + Polio Sabin Group; SB692392 2 dose + Tritanrix + Prevnar + Polio Sabin Group
Biological: Tritanrix™ HB+Hib — Intramuscular, 3 doses
  Arms: Control Tritanrix + Prevnar + Polio Sabin Group; SB692392 1 dose + Tritanrix + Prevnar + Polio Sabin Group; SB692392 2 dose + Tritanrix + Prevnar + Polio Sabin Group
Biological: Prevnar™ — Intramuscular, 3 doses
  Arms: Control Tritanrix + Prevnar + Polio Sabin Group; SB692392 1 dose + Tritanrix + Prevnar + Polio Sabin Group; SB692392 2 dose + Tritanrix + Prevnar + Polio Sabin Group
Biological: Polio Sabin™ — Oral, 3 doses
  Arms: Control Tritanrix + Prevnar + Polio Sabin Group; SB692392 1 dose + Tritanrix + Prevnar + Polio Sabin Group; SB692392 2 dose + Tritanrix + Prevnar + Polio Sabin Group
Biological: Menjugate™ — Intramuscular, 3 doses
  Arms: Control Menjugate Group

SUMMARY:
This purpose of the study is to assess the safety and immunogenicity of a GSK Biologicals' candidate tuberculosis vaccine (692342) when administered concomitantly with or after the Expanded Programme of Immunisation vaccines regimen to healthy infants aged between and including 2 and 7 months, living in a tuberculosis endemic region.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects who the investigator believes that their parent(s)/ Legally Acceptable Representative (LAR(s)) can and will comply with the requirements of the protocol.
* Written or oral, signed or thumb-printed and witnessed informed consent obtained from the subject's parent(s)/LAR(s).
* Subjects who received their birth dose of Bacille Calmette Guerrin.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

For the 'Outside Expanded Programme on Immunisation' cohort:

* Must have documented evidence that he/she has completed the primary Expanded Programme on Immunisation regimen at least 1 month prior to planned vaccination with investigational vaccination regimen.
* Aged between 5 and 7 months at the time of the first study vaccination.

For the 'Within EPI' cohort:

* Must have received the birth dose of Bacille Calmette Guerrin, oral polio vaccine and Hepatitis B vaccine but NO further Expanded Programme on Immunisation vaccines.
* Aged between 2 and 4 months at the time of the first study vaccination with diphtheria, tetanus, whole cell pertussis/ Haemophilus influenzae type b vaccine + pneumococcal conjugate vaccine + oral polio vaccine.

Exclusion Criteria:

* Child in care
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal abnormality, as determined by physical examination and/or laboratory screening tests.
* Laboratory screening tests out of range, which in the investigator's opinion affects the ability of the child to take part in the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency.
* Major congenital defects.
* History of any neurological disorders or seizures.
* Any condition or illness or medication, which in the opinion of the investigator might interfere with the evaluation of the safety or immunogenicity of the study vaccine.
* Any other findings that the investigator feels would increase the risk of having an adverse outcome from participation in the trial.
* Acute disease and/or fever at the time of enrolment.
* Use of any investigational or non-registered product other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* For the 'Within Expanded Programme on Immunisation' Cohort only: Previous vaccination with diphtheria, tetanus, pertussis, Haemophilus influenzae type b and pneumococcal conjugate vaccine.
* History of previous administration of experimental Mycobacterium tuberculosis vaccines.
* Administration of immunoglobulins, blood transfusions and/or other blood products since birth to the first dose of study vaccine or planned administration during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned participation or concurrently participating in another clinical study at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Any chronic drug therapy to be continued during the study period, with the exception of vitamins and/or dietary supplements
* History of allergic reactions or anaphylaxis to any vaccine.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study vaccines.
* Severe malnutrition at screening defined as weight-for-age Z-score < -3 standard deviation.
* Children will not be enrolled if any maternal, obstetrical or neonatal event that has occurred might, in the judgment of the investigator, result in increased neonatal/infant morbidity.

Ages: 2 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 301 (Actual)
Dates: Start 2010-07-07 (Actual); Primary Completion 2011-04-30 (Actual); Study Completion 2012-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Idoko OT, Owolabi OA, Owiafe PK, Moris P, Odutola A, Bollaerts A, Ogundare E, Jongert E, Demoitie MA, Ofori-Anyinam O, Ota MO. Safety and immunogenicity of the M72/AS01 candidate tuberculosis vaccine when given as a booster to BCG in Gambian infants: an open-label randomized controlled trial. Tuberculosis (Edinb). 2014 Dec;94(6):564-78. doi: 10.1016/j.tube.2014.07.001. Epub 2014 Aug 9. PMID 25305000

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One enrolled subject was not administered any vaccine and hence was not considered as having started the study.
Period: Active Phase
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Started | 50 | 50 | 50 | 49 | 52 | 49
Completed | 48 | 49 | 45 | 49 | 52 | 49
Not Completed | 2 | 1 | 5 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Period: Follow Up Phase
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Started | 48 | 49 | 45 | 49 | 52 | 49
Completed | 48 | 49 | 45 | 47 | 50 | 44
Not Completed | 0 | 0 | 0 | 2 | 2 | 5
Not completed — Travelled out of study area | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group | Total
Number analyzed (Participants) | 50 | 50 | 50 | 49 | 52 | 49 | 300
Age, Continuous [Mean (Standard Deviation); unit: Months] | 5.8 (0.68) | 5.7 (0.61) | 5.7 (0.65) | 2.1 (0.28) | 2 (0.19) | 2.1 (0.31) | 3.9 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 20 | 23 | 25 | 16 | 23 | 141
  Male | 16 | 30 | 27 | 24 | 36 | 26 | 159
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 50 | 50 | 50 | 49 | 52 | 49 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3 Solicited Local Symptoms After Dose 1, Dose 2 and Across Doses
Description: Solicited local symptoms assessed were pain, redness and swelling. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: From Day 0 to Day 6
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects for whom data were available. As the outcome was defined differently according to the doses received by the subjects in each group, it is presented separately.
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Grade 3 Pain, Dose 1 | 0 | 0 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 49 | 0 | 48
  Grade 3 Pain, Dose 2 | 0 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 49 | 0 | 48
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0
  Grade 3 Pain, Across doses | 0 | 0 | 0
  Grade 3 Swelling, Across doses | 0 | 0 | 0

2. Primary Outcome: Number of Subjects With Grade 3 Solicited Local Symptoms After Dose 2, Dose 3 and Across Doses.
Description: Solicited local symptoms were only collected after Dose 2 of EPI vaccination. Solicited local symptoms assessed were pain, redness and swelling. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 20 millimeters (mm) of injection site.
Time Frame: From Day 0 to Day 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 47 | 52 | 48
Participants
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 47 | 0 | 47
  Grade 3 Pain, Dose 2 | 0 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 47 | 0 | 47
  Grade 3 Swelling, Dose 2 | 2 | 0 | 2
  Grade 3 Pain, Dose 3 | 2 | 0 | 0
  Grade 3 Swelling, Dose 3 | 3 | 6 | 3
  Grade 3 Pain, Across doses | 2 | 0 | 0
  Grade 3 Swelling, Across doses | 3 | 6 | 5

3. Primary Outcome: Number of Subjects With Grade 3 Solicited General Symptoms After Dose 1, Dose 2 and Across Doses.
Description: Solicited general symptoms assessed were drowsiness, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], irritability/fussiness and loss of appetite. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C.
Time Frame: From Day 0 to Day 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Grade 3 Drowsiness, Dose 1 | 0 | 0 | 0
  Grade 3 Irritability, Dose 1 | 0 | 0 | 0
  Grade 3 Loss of appetite, Dose 1 | 0 | 0 | 0
  Grade 3 Temperature /Axillary, Dose 1 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 49 | 0 | 48
  Grade 3 Drowsiness, Dose 2 | 0 | 0 | 0
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 49 | 0 | 48
  Grade 3 Irritability, Dose 2 | 0 | 0 | 0
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 49 | 0 | 48
  Grade 3 Loss of appetite, Dose 2 | 0 | 0 | 0
  Grade 3 Temperature/Axillary, Dose 2: number analyzed (Participants) | 49 | 0 | 48
  Grade 3 Temperature/Axillary, Dose 2 | 0 | 0 | 1
  Grade 3 Drowsiness, Across doses | 0 | 0 | 0
  Grade 3 Irritability, Across doses | 0 | 0 | 0
  Grade 3 Loss of appetite, Across doses | 0 | 0 | 0
  Grade 3 Temperature/Axillary, Across doses | 0 | 0 | 1

4. Primary Outcome: Number of Subjects With Grade 3 Solicited General Symptoms After Dose 2, Dose 3 and Across Doses.
Description: Solicited general symptoms were only collected after Dose 2 of EPI vaccination. Solicited general symptoms assessed were drowsiness, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], irritability/fussiness and loss of appetite. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.0 °C.
Time Frame: From Day 0 to Day 6
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 47 | 52 | 48
Participants
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 47 | 0 | 47
  Grade 3 Drowsiness, Dose 2 | 0 | 0 | 0
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 47 | 0 | 47
  Grade 3 Irritability, Dose 2 | 0 | 0 | 0
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 47 | 0 | 47
  Grade 3 Loss of appetite, Dose 2 | 0 | 0 | 0
  Grade 3 Temperature/Axillary, Dose 2: number analyzed (Participants) | 47 | 0 | 47
  Grade 3 Temperature/Axillary, Dose 2 | 0 | 0 | 0
  Grade 3 Drowsiness, Dose 3 | 0 | 0 | 0
  Grade 3 Irritability, Dose 3 | 2 | 0 | 0
  Grade 3 Loss of appetite, Dose 3 | 0 | 0 | 0
  Grade 3 Temperature/Axillary, Dose 3 | 0 | 0 | 0
  Grade 3 Drowsiness, Across doses | 0 | 0 | 0
  Grade 3 Irritability, Across doses | 2 | 0 | 0
  Grade 3 Loss of appetite, Across doses | 0 | 0 | 0
  Grade 3 Temperature/Axillary, Across doses | 0 | 0 | 0

5. Primary Outcome: Number of Subjects With Grade 3 Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: From Day 0 to Day 29
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 50 | 47 | 50 | 52 | 50 | 48
Participants | 28 | 25 | 27 | 14 | 26 | 22

6. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 to Month 17
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 49
Participants | 0 | 1 | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: Haematological/Biochemical parameters assessed were: Haemoglobin (Haem), White Blood Cells (WBC), Platelets (PLA), Alanine Aminotransferase (ALA) and Creatinine (CREA). Grade 3 = Haem.: < 5.0 grams per deciliter (g/dL); WBC.: 1.0 to 1.4 x 10³/micro liter (µL); PLA.: < 25x10³/µL; ALA.: 5.1 to 10.0 x upper limit of normal (ULN) and CREA: 3.1 to 6.0 x ULN.
Time Frame: At Day 0
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 49
Participants
  Haem, PRE, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, PRE, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, PRE, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  ALA, PRE, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, PRE, Grade 3 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: Haematological/Biochemical parameters assessed were: Haemoglobin (Haem), White Blood Cells (WBC), Platelets (PLA), Alanine Aminotransferase (ALA) and Creatinine (CREA). Grade 3 = Haem.: < 5.0 g/dL; WBC.: 1.0 to 1.4 x 10³/µL; PLA.: < 25x10³/µL; ALA.: 5.1 to 10.0 x ULN and CREA: 3.1 to 6.0 x ULN.
Time Frame: At Day 7
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects for whom data were available. Arms were presented separately due to the different timepoints used for reporting the results.
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Haem Grade 3 | 0 | 0 | 0
  WBC Grade 3 | 0 | 0 | 0
  PLA Grade 3 | 0 | 0 | 0
  ALA Grade 3 | 0 | 0 | 0
  CREA Grade 3 | 0 | 0 | 0

9. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Day 37
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 50 | 49 | 52 | 50 | 49
Participants
  Haem Grade 3 | 0 | 0 | 0 | 0 | 0
  WBC Grade 3 | 0 | 0 | 0 | 0 | 0
  PLA Grade 3 | 0 | 0 | 0 | 0 | 0
  ALA Grade 3 | 0 | 0 | 0 | 0 | 0
  CREA Grade 3 | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Day 67
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 49 | 52 | 49
Participants
  Haem Grade 3 | 0 | 0 | 0
  WBC Grade 3 | 0 | 0 | 0
  PLA Grade 3 | 0 | 0 | 0
  ALA Grade 3 | 0 | 0 | 0
  CREA Grade 3 | 0 | 0 | 0

11. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Month 1
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Haem Grade 3 | 0 | 0 | 0
  WBC Grade 3 | 0 | 0 | 0
  PLA Grade 3 | 0 | 0 | 0
  ALA Grade 3 | 0 | 0 | 0
  CREA Grade 3 | 0 | 0 | 0

12. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Month 2
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50
Participants
  Haem Grade 3 | 0 | 0
  WBC Grade 3 | 0 | 0
  PLA Grade 3 | 0 | 0
  ALA Grade 3 | 0 | 0
  CREA Grade 3 | 0 | 0

13. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Month 3
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 49 | 52 | 49
Participants
  Haem Grade 3 | 0 | 0 | 0
  WBC Grade 3 | 0 | 0 | 0
  PLA Grade 3 | 0 | 0 | 0
  ALA Grade 3 | 0 | 0 | 0
  CREA Grade 3 | 0 | 0 | 0

14. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: Haematological/Biochemical parameters assessed were: Haemoglobin (Haem), White Blood Cells (WBC), Platelets (PLA), Alanine Aminotransferase (ALA) and Creatinine (CREA).Grade 3 = Haem.: < 5.0 g/dL; WBC.: 1.0 to 1.4 x 10³/µL; PLA.: < 25x10³/µL; ALA.: 5.1 to 10.0 x ULN and CREA: 3.1 to 6.0 x ULN.
Time Frame: At Month 6
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 1 Dose Group
Number analyzed (Participants) | 50
Participants
  Haem Grade 3 | 0
  WBC Grade 3 | 0
  PLA Grade 3 | 0
  ALA Grade 3 | 0
  CREA Grade 3 | 0

15. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Month 7
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50
Participants
  Haem Grade 3 | 0 | 0
  WBC Grade 3 | 0 | 0
  PLA Grade 3 | 0 | 0
  ALA Grade 3 | 0 | 0
  CREA Grade 3 | 0 | 0

16. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: Six Months post Dose 3 [At Month 13]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50
Participants
  Haem Grade 3 | 0 | 0
  WBC Grade 3 | 0 | 0
  PLA Grade 3 | 0 | 0
  ALA Grade 3 | 0 | 0
  CREA Grade 3 | 0 | 0

17. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Month 12
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group
Number analyzed (Participants) | 50
Participants
  Haem Grade 3 | 0
  WBC Grade 3 | 0
  PLA Grade 3 | 0
  ALA Grade 3 | 0
  CREA Grade 3 | 0

18. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: Twelve Months post Dose 2 [At Month 13]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50
Participants
  Haem Grade 3 | 0 | 0
  WBC Grade 3 | 0 | 0
  PLA Grade 3 | 0 | 0
  ALA Grade 3 | 0 | 0
  CREA Grade 3 | 0 | 0

19. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Month 14
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 49 | 52 | 49
Participants
  Haem Grade 3 | 0 | 0 | 0
  WBC Grade 3 | 0 | 0 | 0
  PLA Grade 3 | 0 | 0 | 1
  ALA Grade 3 | 0 | 0 | 0
  CREA Grade 3 | 0 | 0 | 0

20. Primary Outcome: Number of Subjects With Grade 3 Haematological and Biochemical Levels
Description: as for outcome 8
Time Frame: At Month 8
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 49 | 50 | 49
Participants
  Haem Grade 3 | 0 | 0 | 0
  WBC Grade 3 | 0 | 0 | 0
  PLA Grade 3 | 0 | 0 | 0
  ALA Grade 3 | 0 | 1 | 0
  CREA Grade 3 | 0 | 0 | 0

21. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)4+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: Immune markers expressed were among Interleukin-2 (IL-2),Interferon-gamma (INF-γ),Tumour necrosis factor-alpha (TNF-α) and CD40-ligand (CD40-L).
Time Frame: Before vaccination (PRE)
Population: The analysis was performed on the ATP cohort for analysis of immunogenicity which included all evaluable subjects (i.e., those meeting all eligibility criteria, complying with the procedures defined in the protocol, with no elimination criteria during the study), for whom data concerning immunogenicity outcome measures were available.
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 37 | 36 | 42 | 39 | 34 | 39
T cells/million cells
  CD4 all doubles, PRE | 47 [23 to 87] | 59.5 [30.5 to 125] | 42.5 [22 to 71] | 88 [27 to 181] | 44.5 [11 to 65] | 52 [33 to 149]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), PRE | 1 [1 to 1] | 1 [1 to 24.5] | 1 [1 to 12] | 14 [1 to 53] | 1 [1 to 15] | 1 [1 to 30]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-), PRE | 1 [1 to 12] | 1 [1 to 12] | 1 [1 to 1] | 1 [1 to 17] | 1 [1 to 1] | 1 [1 to 14]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+), PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-), PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+), PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-), PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+), PRE | 1 [1 to 11] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 15] | 1 [1 to 1] | 1 [1 to 13]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-), PRE | 14 [1 to 51] | 1 [1 to 28] | 11.5 [1 to 41] | 3 [1 to 62] | 1 [1 to 16] | 1 [1 to 52]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+), PRE | 1 [1 to 12] | 1 [1 to 24] | 1 [1 to 12] | 1 [1 to 27] | 1 [1 to 1] | 1 [1 to 27]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-), PRE | 1 [1 to 12] | 1 [1 to 6] | 1 [1 to 12] | 1 [1 to 1] | 1 [1 to 11] | 1 [1 to 16]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+), PRE | 1 [1 to 1] | 1 [1 to 11.5] | 1 [1 to 1] | 1 [1 to 20] | 1 [1 to 1] | 1 [1 to 15]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-), PRE | 1 [1 to 38] | 5.5 [1 to 29.5] | 1 [1 to 40] | 28 [1 to 63] | 1 [1 to 40] | 20 [1 to 62]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+), PRE | 1 [1 to 1] | 1 [1 to 12.5] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-), PRE | 1 [1 to 11] | 1 [1 to 27.5] | 1 [1 to 19] | 1 [1 to 11] | 1.5 [1 to 14] | 1 [1 to 21]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+), PRE | 1 [1 to 11] | 1 [1 to 21.5] | 1 [1 to 13] | 12 [1 to 47] | 1 [1 to 22] | 15 [1 to 49]

22. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)4+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: Immune markers expressed were among Interleukin-2 (IL-2) and/or Interferon-gamma (INF-γ) and/or Tumour necrosis factor-alpha (TNF-α) and/or CD40-ligand (CD40-L).
Time Frame: Seven Days post each dose (D7)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 37 | 42 | 43 | 43 | 37 | 44
T cells/million cells
  CD4 all doubles, D7 | 499 [250 to 1267] | 593.5 [269 to 1094] | 128 [83 to 379] | 174 [67 to 321] | 55 [33 to 81] | 52.5 [33 to 85]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), D7 | 24 [1 to 83] | 42.5 [14 to 66] | 1 [1 to 39] | 16 [1 to 43] | 1 [1 to 15] | 1 [1 to 19]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-), D7 | 47 [15 to 143] | 61.5 [18 to 157] | 12 [1 to 25] | 12 [1 to 29] | 1 [1 to 12] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+), D7 | 25 [1 to 103] | 19.5 [1 to 71] | 1 [1 to 26] | 13 [1 to 38] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-), D7 | 65 [12 to 286] | 82.5 [29 to 320] | 24 [1 to 52] | 14 [1 to 44] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+), D7 | 1 [1 to 15] | 1 [1 to 22] | 1 [1 to 1] | 1 [1 to 12] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-), D7 | 1 [1 to 32] | 11 [1 to 38] | 1 [1 to 11] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+), D7 | 19 [9 to 61] | 36.5 [1 to 105] | 1 [1 to 19] | 13 [1 to 49] | 1 [1 to 1] | 1 [1 to 13]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-), D7 | 52 [1 to 144] | 112 [25 to 297] | 24 [1 to 102] | 21 [1 to 58] | 9 [1 to 63] | 1 [1 to 37]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+), D7 | 12 [1 to 32] | 14.5 [1 to 45] | 1 [1 to 24] | 1 [1 to 21] | 1 [1 to 12] | 11.5 [1 to 15.5]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-), D7 | 64 [12 to 107] | 35.5 [1 to 88] | 3 [1 to 24] | 1 [1 to 13] | 1 [1 to 13] | 1 [1 to 7.5]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+), D7 | 173 [38 to 232] | 102 [31 to 237] | 22 [1 to 86] | 22 [1 to 67] | 1 [1 to 1] | 1 [1 to 14.5]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-), D7 | 576 [245 to 1126] | 493 [309 to 960] | 138 [42 to 208] | 26 [1 to 134] | 1 [1 to 45] | 1 [1 to 42.5]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+), D7 | 1 [1 to 18] | 1 [1 to 36] | 1 [1 to 11] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-), D7 | 25 [10 to 58] | 27.5 [5 to 85] | 1 [1 to 28] | 1 [1 to 20] | 11 [1 to 21] | 1 [1 to 13.5]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+), D7 | 232 [85 to 444] | 160.5 [61 to 314] | 30 [5 to 69] | 40 [12 to 91] | 1 [1 to 17] | 14 [1 to 44.5]

23. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)4+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: as for outcome 22
Time Frame: One Month post each dose (M1)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 41 | 43 | 44 | 41 | 34 | 42
T cells/million cells
  CD4 all doubles, M1 | 640 [403 to 1200] | 859 [348 to 1950] | 173.5 [93.5 to 476] | 235 [142 to 485] | 31 [22 to 66] | 55.5 [30 to 115]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), M1 | 52 [1 to 157] | 50 [12 to 253] | 17 [1 to 63] | 25 [1 to 88] | 1 [1 to 12] | 12 [1 to 26]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-), M1 | 142 [48 to 300] | 195 [66 to 408] | 30 [11.5 to 82.5] | 56 [14 to 88] | 1 [1 to 12] | 1 [1 to 17]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+), M1 | 14 [1 to 45] | 24 [1 to 132] | 1 [1 to 14] | 12 [1 to 26] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-), M1 | 109 [49 to 143] | 138 [56 to 327] | 27 [1 to 59] | 28 [12 to 63] | 1 [1 to 1] | 1 [1 to 12]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+), M1 | 1 [1 to 19] | 17 [1 to 37] | 1 [1 to 1] | 1 [1 to 12] | 1 [1 to 1] | 1 [1 to 11]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-), M1 | 15 [1 to 44] | 14 [1 to 63] | 1 [1 to 6] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 12]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+), M1 | 14 [1 to 41] | 24 [1 to 64] | 1 [1 to 12] | 12 [1 to 24] | 1 [1 to 1] | 1 [1 to 14]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-), M1 | 51 [1 to 107] | 51 [1 to 162] | 1 [1 to 50.5] | 16 [1 to 96] | 1 [1 to 42] | 1 [1 to 42]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+), M1 | 28 [1 to 109] | 20 [1 to 60] | 1 [1 to 45] | 12 [1 to 24] | 1 [1 to 1] | 1 [1 to 15]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-), M1 | 95 [32 to 251] | 127 [63 to 257] | 28 [1 to 59.5] | 15 [1 to 78] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+), M1 | 57 [26 to 204] | 63 [27 to 118] | 19 [1 to 76] | 24 [1 to 44] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-), M1 | 431 [239 to 838] | 449 [253 to 793] | 115.5 [42.5 to 277.5] | 127 [36 to 257] | 3 [1 to 33] | 23 [1 to 66]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+), M1 | 1 [1 to 27] | 1 [1 to 29] | 1 [1 to 7] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-), M1 | 53 [5 to 106] | 51 [3 to 108] | 9.5 [1 to 38] | 19 [1 to 58] | 1 [1 to 15] | 11 [1 to 35]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+), M1 | 54 [18 to 107] | 71 [25 to 141] | 19.5 [1 to 49] | 11 [1 to 48] | 1 [1 to 14] | 1 [1 to 21]

24. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)4+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: as for outcome 22
Time Frame: Six Months post each dose (M6)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 36 | 40 | 42 | 43 | 34 | 44
T cells/million cells
  CD4 all doubles, M6 | 633 [324 to 1062] | 512 [318.5 to 992.5] | 107.5 [47 to 184] | 107 [72 to 191] | 39 [23 to 71] | 41 [23 to 73.5]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), M6 | 63 [18.5 to 129] | 65 [13 to 125] | 12 [1 to 28] | 16 [1 to 48] | 1 [1 to 13] | 1 [1 to 13.5]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-), M6 | 223 [78 to 403] | 202.5 [101.5 to 434] | 28 [1 to 50] | 17 [1 to 64] | 1 [1 to 15] | 1 [1 to 12.5]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+), M6 | 18.5 [1 to 25.5] | 15.5 [1 to 29] | 1 [1 to 1] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-), M6 | 68.5 [40.5 to 163] | 65 [34.5 to 184.5] | 1 [1 to 22] | 13 [1 to 41] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+), M6 | 1 [1 to 1] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-), M6 | 12 [1 to 20.5] | 1 [1 to 26] | 1 [1 to 11] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+), M6 | 1 [1 to 6.5] | 1 [1 to 28] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 11] | 1 [1 to 13]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-), M6 | 16.5 [1 to 71] | 40.5 [1 to 95.5] | 1 [1 to 28] | 2 [1 to 44] | 1 [1 to 39] | 13.5 [1 to 48.5]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+), M6 | 13.5 [1 to 59.5] | 13 [1 to 52.5] | 1 [1 to 14] | 1 [1 to 17] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-), M6 | 72 [38 to 206.5] | 86.5 [27 to 156.5] | 12 [1 to 28] | 5 [1 to 40] | 1 [1 to 13] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+), M6 | 31 [1 to 84.5] | 26 [7 to 55] | 1 [1 to 13] | 1 [1 to 16] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-), M6 | 310.5 [60 to 591.5] | 171.5 [126.5 to 369] | 35.5 [1 to 68] | 48 [8 to 99] | 10 [1 to 27] | 12.5 [1 to 41]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+), M6 | 1 [1 to 18] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-), M6 | 19 [1 to 71.5] | 27 [1 to 61] | 1 [1 to 12] | 1 [1 to 14] | 1 [1 to 14] | 1 [1 to 13.5]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+), M6 | 19.5 [1 to 58] | 14 [1 to 46.5] | 1 [1 to 14] | 1 [1 to 16] | 1 [1 to 18] | 1 [1 to 14]

25. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)4+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: as for outcome 22
Time Frame: Twelve Months post each dose (M12)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 38 | 41 | 45 | 41 | 33 | 43
T cells/million cells
  CD4 all doubles, M12 | 456.5 [237 to 1062] | 403 [245 to 745] | 104 [59 to 201] | 98 [52 to 157] | 38 [22 to 61] | 41 [22 to 79]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), M12 | 51 [18 to 145] | 65 [18 to 99] | 16 [1 to 42] | 14 [1 to 48] | 1 [1 to 1] | 1 [1 to 14]
  CD4.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-), M12 | 176 [73 to 424] | 144 [80 to 329] | 28 [12 to 52] | 26 [13 to 47] | 1 [1 to 14] | 1 [1 to 12]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+), M12 | 7 [1 to 39] | 13 [1 to 40] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-), M12 | 56.5 [24 to 145] | 67 [24 to 149] | 13 [1 to 21] | 1 [1 to 16] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+), M12 | 1 [1 to 13] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-), M12 | 12.5 [1 to 37] | 1 [1 to 23] | 1 [1 to 1] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 12]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+), M12 | 1 [1 to 12] | 1 [1 to 17] | 1 [1 to 13] | 1 [1 to 1] | 1 [1 to 12] | 1 [1 to 13]
  CD4.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-), M12 | 10.5 [1 to 57] | 29 [1 to 81] | 1 [1 to 48] | 14 [1 to 67] | 22 [1 to 58] | 13 [1 to 72]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+), M12 | 13 [1 to 29] | 1 [1 to 17] | 1 [1 to 16] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-), M12 | 60 [15 to 138] | 39 [13 to 91] | 12 [1 to 21] | 1 [1 to 12] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+), M12 | 21 [1 to 56] | 19 [1 to 40] | 1 [1 to 12] | 1 [1 to 12] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-), M12 | 179 [84 to 283] | 155 [74 to 300] | 30 [1 to 66] | 50 [22 to 87] | 1 [1 to 20] | 3 [1 to 25]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+), M12 | 1 [1 to 15] | 1 [1 to 12] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-), M12 | 3.5 [1 to 38] | 1 [1 to 35] | 3 [1 to 40] | 1 [1 to 39] | 1 [1 to 27] | 1 [1 to 19]
  CD4.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+), M12 | 14.5 [1 to 49] | 2 [1 to 54] | 1 [1 to 25] | 1 [1 to 25] | 1 [1 to 27] | 1 [1 to 41]

26. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)8+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: as for outcome 22
Time Frame: Before vaccination (PRE)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 37 | 36 | 42 | 39 | 34 | 39
T cells/million cells
  CD8 all doubles, PRE | 11 [11 to 81] | 40.5 [11 to 70.5] | 11 [11 to 61] | 11 [11 to 93] | 11 [11 to 65] | 11 [11 to 47]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-),PRE | 1 [1 to 44] | 1 [1 to 42] | 1 [1 to 53] | 1 [1 to 46] | 1 [1 to 50] | 1 [1 to 55]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-),PRE | 8 [1 to 116] | 117 [40 to 260] | 57 [1 to 138] | 61 [1 to 166] | 53.5 [1 to 91] | 65 [1 to 302]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+),PRE | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-),PRE | 1 [1 to 64] | 1 [1 to 14.5] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 28] | 1 [1 to 27]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+),PRE | 1 [1 to 40] | 1 [1 to 1] | 1 [1 to 23] | 1 [1 to 1] | 1 [1 to 2] | 1 [1 to 43]

27. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)8+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: as for outcome 22
Time Frame: Seven Days after each dose (D7)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 37 | 42 | 43 | 43 | 37 | 44
T cells/million cells
  CD8 all doubles, D7 | 61 [11 to 147] | 55 [11 to 161] | 43 [11 to 101] | 46 [11 to 82] | 11 [11 to 11] | 11 [11 to 28]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-),D7 | 1 [1 to 1] | 1 [1 to 31] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-),D7 | 34 [1 to 104] | 37 [1 to 119] | 6 [1 to 116] | 1 [1 to 100] | 3 [1 to 54] | 1 [1 to 25]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-),D7 | 61 [1 to 185] | 161.5 [1 to 574] | 1 [1 to 107] | 34 [1 to 303] | 1 [1 to 61] | 123 [1 to 289.5]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+),D7 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-),D7 | 6 [1 to 64] | 7.5 [1 to 72] | 1 [1 to 67] | 1 [1 to 10] | 1 [1 to 85] | 1 [1 to 48]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+),D7 | 37 [1 to 89] | 1 [1 to 50] | 1 [1 to 70] | 1 [1 to 31] | 1 [1 to 30] | 1 [1 to 2.5]

28. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)8+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: as for outcome 22
Time Frame: One Month after each dose (M1)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 41 | 43 | 44 | 41 | 34 | 42
T cells/million cells
  CD8 all doubles, M1 | 69 [11 to 145] | 82 [11 to 163] | 29.5 [11 to 80] | 81 [26 to 139] | 11 [11 to 28] | 11 [11 to 53]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), M1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-),M1 | 1 [1 to 1] | 1 [1 to 32] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+),M1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-),M1 | 1 [1 to 1] | 1 [1 to 32] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+),M1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-),M1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+),M1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 56] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-),M1 | 1 [1 to 55] | 1 [1 to 46] | 1 [1 to 52] | 11 [1 to 99] | 2.5 [1 to 85] | 4 [1 to 109]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+),M1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-),M1 | 1 [1 to 12] | 1 [1 to 28] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+),M1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-),M1 | 1 [1 to 139] | 142 [1 to 308] | 2.5 [1 to 116] | 109 [2 to 218] | 1 [1 to 48] | 86 [1 to 330]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+),M1 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-),M1 | 18 [1 to 87] | 12 [1 to 111] | 1 [1 to 50] | 1 [1 to 90] | 1 [1 to 51] | 1 [1 to 35]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+),M1 | 1 [1 to 65] | 1 [1 to 65] | 1 [1 to 5.5] | 1 [1 to 64] | 1 [1 to 5] | 1 [1 to 1]

29. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)8+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: as for outcome 22
Time Frame: Six Months after each dose (M6)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 36 | 40 | 42 | 43 | 34 | 44
T cells/million cells
  CD8 all doubles, M6 | 11 [11 to 53] | 11 [11 to 20] | 11 [11 to 32] | 11 [11 to 11] | 11 [11 to 29] | 11 [11 to 11]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-),M6 | 1 [1 to 25.5] | 2 [1 to 65] | 1 [1 to 44] | 1 [1 to 63] | 1 [1 to 52] | 2 [1 to 59]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-),M6 | 1 [1 to 29.5] | 27.5 [1 to 60] | 38 [1 to 91] | 1 [1 to 56] | 28 [1 to 67] | 1 [1 to 43.5]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+),M6 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-),M6 | 1 [1 to 54.5] | 1 [1 to 55.5] | 1 [1 to 3] | 1 [1 to 60] | 1 [1 to 36] | 1 [1 to 49]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+),M6 | 1 [1 to 33] | 1 [1 to 36.5] | 1 [1 to 1] | 1 [1 to 40] | 1 [1 to 1] | 1 [1 to 1]

30. Secondary Outcome: Frequency of M. Tuberculosis Fusion Protein M72 (M72)-Specific Cluster of Differentiation (CD)8+ T Cells Per Million Cells Expressing at Least Two Different Immune Markers
Description: as for outcome 22
Time Frame: Twelve Months after each dose (M12)
Population: as for outcome 21
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 38 | 41 | 45 | 41 | 33 | 43
T cells/million cells
  CD8 all doubles, M12 | 11 [11 to 52] | 11 [11 to 35] | 11 [11 to 38] | 11 [11 to 41] | 11 [11 to 41] | 11 [11 to 42]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (+), M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α(+)+INF-γ (-),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+INF-γ (+),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(+)+TNF-α (-)+I INF-γ (-),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (+),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α(+)+INF-γ (-),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (+),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(+)+IL-2(-)+TNF-α (-)+INF-γ (-),M12 | 1 [1 to 29] | 1 [1 to 64] | 1 [1 to 68] | 1 [1 to 35] | 1 [1 to 32] | 1 [1 to 40]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (+),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α(+)+INF-γ (-),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (+),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(+)+TNF-α (-)+INF-γ (-),M12 | 14.5 [1 to 92] | 16 [1 to 77] | 1 [1 to 59] | 1 [1 to 35] | 1 [1 to 57] | 15 [1 to 66]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ(+),M12 | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 1] | 1 [1 to 5] | 1 [1 to 1]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (+)+INF-γ (-),M12 | 1 [1 to 34] | 1 [1 to 50] | 1 [1 to 58] | 1 [1 to 65] | 1 [1 to 117] | 1 [1 to 22]
  CD8.CD40-L(-)+IL-2(-)+TNF-α (-)+INF-γ(+),M12 | 1.5 [1 to 67] | 1 [1 to 48] | 1 [1 to 25] | 1 [1 to 128] | 11 [1 to 57] | 1 [1 to 33]

31. Secondary Outcome: Number of Seropositive Subjects Against M72 Antigen
Description: A seropositive subject was a subject whose M72 antibody concentration was greater than or equal to 2.8 ELISA units per millilitre (EL.U/mL).
Time Frame: Before vaccination (PRE) and after each dose [at 1, 6 and 12 months post-vaccination (M1, M6 and M12)]
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 43 | 44 | 48 | 46 | 39 | 46
Participants
  Anti-M72, PRE | 0 | 0 | 0 | 0 | 1 | 0
  Anti-M72, M1: number analyzed (Participants) | 42 | 43 | 45 | 44 | 34 | 43
  Anti-M72, M1 | 42 | 43 | 39 | 39 | 1 | 0
  Anti-M72, M6: number analyzed (Participants) | 40 | 41 | 45 | 45 | 36 | 45
  Anti-M72, M6 | 40 | 41 | 32 | 35 | 0 | 1
  Anti-M72, M12: number analyzed (Participants) | 41 | 42 | 47 | 45 | 35 | 43
  Anti-M72, M12 | 41 | 42 | 35 | 31 | 1 | 2

32. Secondary Outcome: Concentration of Antibodies Against M72 Antigen
Description: Concentrations given in EL.U/mL were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Before vaccination (PRE) and after each dose [at 1, 6 and 12 months post-vaccination (M1, M6 and M12)]
Population: as for outcome 21
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 43 | 44 | 48 | 46 | 39 | 46
EL.U/mL
  Anti-M72, PRE | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.4] | 1.5 [1.3 to 1.7] | 1.4 [1.4 to 1.4]
  Anti-M72, M1: number analyzed (Participants) | 42 | 43 | 45 | 44 | 34 | 43
  Anti-M72, M1 | 1275.2 [981.3 to 1657.2] | 1264 [928 to 1721.5] | 8 [6 to 10.7] | 7.4 [5.3 to 10.2] | 1.5 [1.3 to 1.7] | 1.4 [1.4 to 1.4]
  Anti-M72, M6: number analyzed (Participants) | 40 | 41 | 45 | 45 | 36 | 45
  Anti-M72, M6 | 98.9 [75.2 to 130.1] | 102.6 [78.7 to 133.9] | 4.6 [3.4 to 6.2] | 4.9 [3.8 to 6.4] | 1.4 [1.4 to 1.4] | 1.4 [1.4 to 1.5]
  Anti-M72, M12: number analyzed (Participants) | 41 | 42 | 47 | 45 | 35 | 43
  Anti-M72, M12 | 68.3 [50.7 to 92] | 76 [56.6 to 102] | 5.3 [3.9 to 7] | 4.3 [3.2 to 5.8] | 1.4 [1.4 to 1.5] | 1.5 [1.4 to 1.7]

33. Secondary Outcome: Number of Seroprotected Subjects Against Diphtheria Toxoid (Anti-D) and Tetanus Toxoid (Anti-T)
Description: A seroprotected subject was a subject whose anti-diphtheria toxoid (anti-D)/anti-tetanus toxoid (anti-T) antibody concentration was ≥ 0.1 international-units per millilitre (IU/mL).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: The analysis was performed on those groups from the ATP cohort for analysis of immunogenicity that also contained Tritanrix™ HepB+Hiberix™, Prevnar® and Polio Sabin™ vaccines in their vaccination regimen, which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available.
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 43 | 43 | 43
Participants
  Anti-D, PRE: number analyzed (Participants) | 37 | 38 | 38
  Anti-D, PRE | 6 | 10 | 6
  Anti-D, PIII(M3) | 43 | 43 | 43
  Anti-T, PRE: number analyzed (Participants) | 37 | 38 | 38
  Anti-T, PRE | 32 | 35 | 35
  Anti-T, PIII(M3) | 43 | 43 | 43

34. Secondary Outcome: Anti-D, Anti-T Antibody Concentrations
Description: Concentrations given in IU/mL, were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 43 | 43 | 43
IU/mL
  Anti-D, PRE: number analyzed (Participants) | 37 | 38 | 38
  Anti-D, PRE | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  Anti-D, PIII(M3) | 2.1 [1.6 to 2.7] | 2.4 [1.8 to 3.1] | 2.5 [2 to 3.1]
  Anti-T, PRE: number analyzed (Participants) | 37 | 38 | 38
  Anti-T, PRE | 0.6 [0.4 to 1] | 1 [0.6 to 1.5] | 1 [0.6 to 1.6]
  Anti-T, PIII(M3) | 5.5 [4.3 to 7.1] | 4.8 [3.6 to 6.4] | 6.3 [4.8 to 8.3]

35. Secondary Outcome: Number of Seroprotected Subjects Against Haemophilus Influenzae Type B (Anti-PRP)
Description: A seroprotected subject was a subject whose anti-PRP antibody concentration was ≥ 0.15 micrograms per millilitre (µg/mL).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 47 | 46 | 48
Participants
  Anti-PRP, PRE | 8 | 14 | 12
  Anti-PRP, PIII(M3): number analyzed (Participants) | 44 | 44 | 43
  Anti-PRP, PIII(M3) | 44 | 44 | 43

36. Secondary Outcome: Anti-PRP Antibody Concentrations
Description: Concentrations given in µg/mL were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 47 | 46 | 48
µg/mL
  Anti-PRP, PRE | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.2] | 0.1 [0.1 to 0.2]
  Anti-PRP, PIII(M3): number analyzed (Participants) | 44 | 44 | 43
  Anti-PRP, PIII(M3) | 28.2 [20.3 to 39.1] | 30.3 [21.8 to 42.1] | 31.2 [21.8 to 44.7]

37. Secondary Outcome: Number of Seropositive Subjects Against Bordetella Pertussis (Anti-BPT)
Description: A seropositive subject was a subject whose anti-BPT antibody concentration was ≥ 15 EL.U/mL.
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 44 | 43 | 43
Participants
  Anti-BPT, PRE: number analyzed (Participants) | 41 | 40 | 43
  Anti-BPT, PRE | 1 | 1 | 1
  Anti-BPT, PIII(M3) | 44 | 43 | 43

38. Secondary Outcome: Anti-BPT Antibody Concentrations
Description: Concentrations given in EL.U/mL were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 44 | 43 | 43
EL.U/mL
  Anti-BPT, PRE: number analyzed (Participants) | 41 | 40 | 43
  Anti-BPT, PRE | 7.7 [7.3 to 8] | 7.6 [7.4 to 7.9] | 7.6 [7.4 to 7.9]
  Anti-BPT, PIII(M3) | 139.4 [117.7 to 164.9] | 132.1 [116.6 to 149.5] | 131.5 [113.5 to 152.5]

39. Secondary Outcome: Number of Seropositive Subjects Against Hepatitis B (Anti-HB)
Description: A seropositive subject was a subject whose anti-HB antibody concentration was ≥ 10 milli-international units per millilitre (mIU/mL).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 44 | 44 | 43
Participants
  Anti-HB, PRE: number analyzed (Participants) | 41 | 40 | 41
  Anti-HB, PRE | 9 | 14 | 13
  Anti-HB, PIII(M3) | 42 | 43 | 42

40. Secondary Outcome: Number of Seropositive Subjects Against Hepatitis B (Anti-HB) With Antibody Concentrations ≥100mIU/mL
Description: A decrease in the specificity of the anti-HB ELISA assay had been observed in some studies for low levels of antibody (10-100 mIU/mL). The table shows updated results following partial or complete retesting/reanalysis. Following from this, the table shows data with titers ≥ 100 mIU/mL.
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 44 | 44 | 43
Participants
  Anti-HB, PRE: number analyzed (Participants) | 41 | 40 | 41
  Anti-HB, PRE | 2 | 2 | 2
  Anti-HB, PIII(M3) | 42 | 42 | 42

41. Secondary Outcome: Anti-HB Antibody Concentrations
Description: Concentrations given in mIU/mL were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 44 | 44 | 43
mIU/mL
  Anti-HB, PRE: number analyzed (Participants) | 41 | 40 | 41
  Anti-HB, PRE | 8.3 [6 to 11.4] | 10 [7.1 to 14] | 9 [6.7 to 12.2]
  Anti-HB, PIII(M3) | 1725.5 [1045 to 2849] | 1471.8 [947.5 to 2286] | 2153 [1468.2 to 3157.4]

42. Secondary Outcome: Number of Seropositive Subjects Against Polio (Anti-Polio1, Anti-Polio2, Anti-Polio3)
Description: A seropositive subject was a subject whose anti-polio antibody titer was ≥ 1:8.
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 46 | 45 | 48
Participants
  Anti-Polio1, PRE | 36 | 38 | 39
  Anti-Polio1, PIII(M3): number analyzed (Participants) | 44 | 44 | 43
  Anti-Polio1, PIII(M3) | 41 | 43 | 42
  Anti-Polio2, PRE | 33 | 32 | 38
  Anti-Polio2, PIII(M3): number analyzed (Participants) | 44 | 44 | 43
  Anti-Polio2, PIII(M3) | 43 | 42 | 42
  Anti-Polio3, PRE | 21 | 18 | 14
  Anti-Polio3, PIII(M3): number analyzed (Participants) | 44 | 44 | 43
  Anti-Polio3, PIII(M3) | 42 | 38 | 39

43. Secondary Outcome: Anti-Polio1, Anti-Polio2, Anti-Polio3 Antibody Titers
Description: Concentrations given in titers were expressed as Geometric Mean Titers (GMTs).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 46 | 45 | 48
Titers
  Anti-Polio1, PRE | 56.3 [30.7 to 103.2] | 48.8 [27.3 to 87.5] | 103.8 [58.1 to 185.3]
  Anti-Polio1, PIII(M3): number analyzed (Participants) | 44 | 44 | 43
  Anti-Polio1, PIII(M3) | 299.9 [167.6 to 536.7] | 397.8 [240.2 to 658.8] | 573.1 [368.7 to 890.6]
  Anti-Polio2, PRE | 51.8 [28.8 to 93.2] | 53.2 [28 to 101] | 61.2 [34.8 to 107.8]
  Anti-Polio2, PIII(M3): number analyzed (Participants) | 44 | 44 | 43
  Anti-Polio2, PIII(M3) | 458.7 [307.7 to 683.7] | 524.3 [331.1 to 830.3] | 499.9 [317.7 to 786.5]
  Anti-Polio3, PRE | 15.2 [9 to 25.6] | 15.4 [8.6 to 27.6] | 10.9 [6.7 to 17.9]
  Anti-Polio3, PIII(M3): number analyzed (Participants) | 44 | 44 | 43
  Anti-Polio3, PIII(M3) | 154.8 [100.8 to 237.8] | 103.5 [59.7 to 179.6] | 123 [73.6 to 205.8]

44. Secondary Outcome: Number of Seropositive Subjects Against Streptococcus Pneumoniae (Anti-4, Anti-6B, Anti-9V, Anti-14, Anti-18C, Anti-19F, Anti-23F)
Description: A seropositive subject was a subject whose anti-S pneumoniae antibody concentration was ≥ 0.05 µg/mL.
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 44 | 44 | 43
Participants
  Anti-4, PRE: number analyzed (Participants) | 39 | 39 | 40
  Anti-4, PRE | 18 | 21 | 12
  Anti-4, PIII(M3): number analyzed (Participants) | 43 | 43 | 43
  Anti-4, PIII(M3) | 43 | 43 | 43
  Anti-6B, PRE: number analyzed (Participants) | 38 | 39 | 40
  Anti-6B, PRE | 29 | 27 | 26
  Anti-6B, PIII(M3): number analyzed (Participants) | 44 | 43 | 43
  Anti-6B, PIII(M3) | 44 | 41 | 40
  Anti-9V, PRE: number analyzed (Participants) | 37 | 39 | 39
  Anti-9V, PRE | 28 | 33 | 25
  Anti-9V,PIII(M3): number analyzed (Participants) | 43 | 43 | 43
  Anti-9V,PIII(M3) | 43 | 43 | 43
  Anti-14, PRE: number analyzed (Participants) | 39 | 38 | 40
  Anti-14, PRE | 39 | 38 | 38
  Anti-14, PIII(M3) | 44 | 44 | 43
  Anti-18C, PRE: number analyzed (Participants) | 42 | 40 | 42
  Anti-18C, PRE | 30 | 35 | 26
  Anti-18C, PIII(M3): number analyzed (Participants) | 43 | 44 | 43
  Anti-18C, PIII(M3) | 43 | 44 | 43
  Anti-19F, PRE: number analyzed (Participants) | 37 | 38 | 40
  Anti-19F, PRE | 35 | 37 | 39
  Anti-19F, PIII(M3) | 44 | 44 | 43
  Anti-23F, PRE: number analyzed (Participants) | 41 | 40 | 42
  Anti-23F, PRE | 25 | 30 | 26
  Anti-23F, PIII(M3): number analyzed (Participants) | 44 | 43 | 43
  Anti-23F, PIII(M3) | 43 | 43 | 42

45. Secondary Outcome: Number of Subjects With S. Pneumoniae Antibody Concentrations ≥ 0.2 Microgram/Milliliter
Description: A seroconverted subject is a vaccinated subject with at least a four fold increased antibody titer post vaccination.
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 44 | 44 | 43
Participants
  Anti-4, PRE: number analyzed (Participants) | 39 | 39 | 40
  Anti-4, PRE | 5 | 10 | 2
  Anti-4, PIII(M3): number analyzed (Participants) | 43 | 43 | 43
  Anti-4, PIII(M3) | 43 | 43 | 43
  Anti-6B, PRE: number analyzed (Participants) | 38 | 39 | 40
  Anti-6B, PRE | 8 | 5 | 6
  Anti-6B, PIII(M3): number analyzed (Participants) | 44 | 43 | 43
  Anti-6B, PIII(M3) | 38 | 40 | 35
  Anti-9V, PRE: number analyzed (Participants) | 37 | 39 | 39
  Anti-9V, PRE | 18 | 20 | 10
  Anti-9V, PIII(M3): number analyzed (Participants) | 43 | 43 | 43
  Anti-9V, PIII(M3) | 43 | 43 | 43
  Anti-14, PRE: number analyzed (Participants) | 39 | 38 | 40
  Anti-14, PRE | 34 | 33 | 33
  Anti-14, PIII(M3) | 44 | 43 | 43
  Anti-18C, PRE: number analyzed (Participants) | 42 | 40 | 42
  Anti-18C, PRE | 10 | 17 | 9
  Anti-18C, PIII(M3): number analyzed (Participants) | 43 | 44 | 43
  Anti-18C, PIII(M3) | 43 | 43 | 42
  Anti-19F, PRE: number analyzed (Participants) | 37 | 38 | 40
  Anti-19F, PRE | 30 | 30 | 26
  Anti-19F, PIII(M3) | 43 | 44 | 43
  Anti-23F, PRE: number analyzed (Participants) | 41 | 40 | 42
  Anti-23F, PRE | 9 | 11 | 14
  Anti-23F, PIII(M3): number analyzed (Participants) | 44 | 43 | 43
  Anti-23F, PIII(M3) | 42 | 41 | 42

46. Secondary Outcome: Anti-4, Anti-6B, Anti-9V, Anti-14, Anti-18C, Anti-19F, Anti-23F Antibody Concentrations
Description: Concentrations, given in µg/mL, were expressed as Geometric Mean Concentrations (GMCs).
Time Frame: Before vaccination (PRE) and 1 Month post Dose 3 [PIII(M3)]
Population: as for outcome 33
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 44 | 44 | 43
µg/mL
  Anti-4, PRE: number analyzed (Participants) | 39 | 39 | 40
  Anti-4, PRE | 0.1 [0 to 0.1] | 0.1 [0.1 to 0.1] | 0 [0 to 0]
  Anti-4, PIII(M3): number analyzed (Participants) | 43 | 43 | 43
  Anti-4, PIII(M3) | 7.7 [6.2 to 9.7] | 6.4 [5.3 to 7.8] | 8.1 [6.5 to 10]
  Anti-6B, PRE: number analyzed (Participants) | 38 | 39 | 40
  Anti-6B, PRE | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  Anti-6B, PIII(M3): number analyzed (Participants) | 44 | 43 | 43
  Anti-6B, PIII(M3) | 2.3 [1.4 to 3.8] | 1.5 [0.9 to 2.4] | 1.5 [0.8 to 2.7]
  Anti-9V, PRE: number analyzed (Participants) | 37 | 39 | 39
  Anti-9V, PRE | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.3] | 0.1 [0.1 to 0.1]
  Anti-9V, PIII(M3): number analyzed (Participants) | 43 | 43 | 43
  Anti-9V, PIII(M3) | 5.8 [4.4 to 7.7] | 4.1 [3 to 5.6] | 6 [4.5 to 8.1]
  Anti-14, PRE: number analyzed (Participants) | 39 | 38 | 40
  Anti-14, PRE | 0.8 [0.6 to 1.2] | 1.1 [0.7 to 1.6] | 0.7 [0.4 to 1]
  Anti-14, PIII(M3) | 3.6 [2.5 to 5.3] | 3.3 [2.3 to 4.7] | 4.2 [2.8 to 6.2]
  Anti-18C, PRE: number analyzed (Participants) | 42 | 40 | 42
  Anti-18C, PRE | 0.1 [0.1 to 0.1] | 0.2 [0.1 to 0.2] | 0.1 [0.1 to 0.1]
  Anti-18C, PIII(M3): number analyzed (Participants) | 43 | 44 | 43
  Anti-18C, PIII(M3) | 7.2 [5.7 to 9] | 5.1 [3.8 to 7] | 6.1 [4.2 to 8.8]
  Anti-19F, PRE: number analyzed (Participants) | 37 | 38 | 40
  Anti-19F, PRE | 0.4 [0.3 to 0.6] | 0.5 [0.3 to 0.7] | 0.3 [0.2 to 0.5]
  Anti-19F, PIII(M3) | 5.8 [4.1 to 8.2] | 5.4 [4.2 to 6.9] | 5.9 [4.5 to 7.5]
  Anti-23F, PRE: number analyzed (Participants) | 41 | 40 | 42
  Anti-23F, PRE | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1] | 0.1 [0.1 to 0.1]
  Anti-23F, PIII(M3): number analyzed (Participants) | 44 | 43 | 43
  Anti-23F, PIII(M3) | 3.2 [2.1 to 4.8] | 3 [2 to 4.6] | 3.8 [2.5 to 5.7]

47. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 6
Time Frame: From Day 0 up to 12 months post last vaccination
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 49
Participants | 2 | 1 | 3 | 1 | 3 | 1

48. Secondary Outcome: Number of Subjects With Normal, Grade 1 (G1), Grade 2 (G2) or Grade 4 (G4) Haematological and Biochemical Markers
Description: Levels assessed for Haemoglobin (Haem), White Blood Cells (WBC), Platelets (PLA), Alanine Aminotransferase (ALA) and Creatinine (CREA) were: normal, G1, G2 and G4 . Values that did not fall under normal levels or assessed grades were missing.
Time Frame: Before vaccination (PRE)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692342 1 Dose Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 50 | 49 | 50 | 52 | 50 | 49
Participants
  Haem, PRE, Normal | 49 | 48 | 50 | 51 | 48 | 49
  Haem, PRE, G1 | 0 | 1 | 0 | 0 | 1 | 0
  Haem, PRE, G2 | 1 | 0 | 0 | 1 | 0 | 0
  Haem, PRE, G4 | 0 | 0 | 0 | 0 | 0 | 0
  Haem, PRE, Missing | 0 | 0 | 0 | 0 | 1 | 0
  WBC, PRE, Normal | 45 | 48 | 49 | 52 | 43 | 47
  WBC, PRE, G1 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, PRE, G2 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, PRE, G4 | 0 | 0 | 0 | 0 | 0 | 0
  WBC, PRE, Missing | 5 | 1 | 1 | 0 | 7 | 2
  PLA, PRE, Normal | 48 | 49 | 49 | 52 | 48 | 49
  PLA, PRE, G1 | 2 | 0 | 0 | 0 | 1 | 0
  PLA, PRE, G2 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, PRE, G4 | 0 | 0 | 0 | 0 | 0 | 0
  PLA, PRE, Missing | 0 | 0 | 0 | 0 | 1 | 0
  ALA, PRE, Normal | 42 | 47 | 39 | 51 | 40 | 48
  ALA, PRE, G1 | 0 | 1 | 0 | 0 | 0 | 1
  ALA, PRE, G2 | 0 | 0 | 0 | 0 | 1 | 0
  ALA, PRE, G4 | 0 | 0 | 0 | 0 | 0 | 0
  ALA, PRE, Missing | 8 | 1 | 11 | 1 | 9 | 0
  CREA, PRE, Normal | 42 | 48 | 39 | 51 | 41 | 49
  CREA, PRE, G1 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, PRE, G2 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, PRE, G4 | 0 | 0 | 0 | 0 | 0 | 0
  CREA, PRE, Missing | 8 | 1 | 11 | 1 | 9 | 0

49. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: Levels assessed for Haemoglobin (Haem), White Blood Cells (WBC), Platelets (PLA), Alanine Aminotransferase (ALA) and Creatinine (CREA) were : normal, grade 1 (G1), grade 2 (G2) and grade 4 (G4). Values that did not fall under normal levels or assessed grades were missing.
Time Frame: Seven days post Dose 1 [PI(D7)]
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Haem, PI(D7), Normal | 49 | 48 | 48
  Haem, PI(D7), G1 | 0 | 0 | 0
  Haem, PI(D7), G2 | 0 | 0 | 0
  Haem, PI(D7), G4 | 0 | 0 | 0
  Haem, PI(D7), Missing | 1 | 2 | 0
  WBC, PI(D7), Normal | 46 | 47 | 45
  WBC, PI(D7), G1 | 0 | 0 | 0
  WBC, PI(D7), G2 | 0 | 0 | 0
  WBC, PI(D7), G4 | 0 | 0 | 0
  WBC, PI(D7), Missing | 4 | 3 | 5
  PLA, PI(D7), Normal | 49 | 49 | 47
  PLA, PI(D7), G1 | 0 | 1 | 1
  PLA, PI(D7), G2 | 0 | 0 | 0
  PLA, PI(D7), G4 | 0 | 0 | 0
  PLA, PI(D7), Missing | 0 | 0 | 1
  ALA, PI(D7), Normal | 48 | 48 | 48
  ALA, PI(D7), G1 | 0 | 0 | 0
  ALA, PI(D7), G2 | 0 | 0 | 0
  ALA, PI(D7), G4 | 0 | 0 | 0
  ALA, PI(D7), Missing | 2 | 2 | 2
  CREA, PI(D7), Normal | 48 | 48 | 49
  CREA, PI(D7), G1 | 0 | 0 | 0
  CREA, PI(D7), G2 | 0 | 0 | 0
  CREA, PI(D7), G4 | 0 | 0 | 0
  CREA, PI(D7), Missing | 2 | 2 | 1

50. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: Levels assessed for Haemoglobin (Haem), White Blood Cells (WBC), Platelets (PLA), Alanine Aminotransferase (ALA) and Creatinine (CREA) were: normal, grade 1 (G1), grade 2 (G2) and grade 4 (G4). Values that did not fall under normal levels or assessed grades were missing.
Time Frame: Seven days post Dose 2 [PII(D37)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Menjugate Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 50 | 49 | 52 | 50 | 49
Participants
  Haem, PII(D37), Normal | 47 | 45 | 0 | 47 | 47
  Haem, PII(D37), G1 | 1 | 0 | 0 | 1 | 0
  Haem, PII(D37), G2 | 0 | 0 | 0 | 0 | 0
  Haem, PII(D37), G4 | 0 | 0 | 0 | 0 | 0
  Haem, PII(D37), Missing | 2 | 4 | 52 | 2 | 2
  WBC, PII(D37), Normal | 42 | 44 | 0 | 44 | 44
  WBC, PII(D37), G1 | 0 | 0 | 0 | 0 | 0
  WBC, PII(D37), G2 | 0 | 0 | 0 | 0 | 0
  WBC, PII(D37), G4 | 0 | 0 | 0 | 0 | 0
  WBC, PII(D37), Missing | 8 | 5 | 52 | 6 | 5
  PLA, PII(D37), Normal | 47 | 45 | 0 | 48 | 47
  PLA, PII(D37), G1 | 1 | 0 | 0 | 0 | 0
  PLA, PII(D37), G2 | 0 | 0 | 0 | 0 | 0
  PLA, PII(D37), G4 | 0 | 0 | 0 | 0 | 0
  PLA, PII(D37), Missing | 2 | 4 | 52 | 2 | 2
  ALA, PII(D37), Normal | 48 | 46 | 0 | 48 | 47
  ALA, PII(D37), G1 | 0 | 0 | 0 | 0 | 0
  ALA, PII(D37), G2 | 0 | 0 | 0 | 0 | 0
  ALA, PII(D37), G4 | 0 | 0 | 0 | 0 | 0
  ALA, PII(D37), Missing | 2 | 3 | 52 | 2 | 2
  CREA, PII(D37), Normal | 48 | 46 | 0 | 48 | 47
  CREA, PII(D37), G1 | 0 | 0 | 0 | 0 | 0
  CREA, PII(D37), G2 | 0 | 0 | 0 | 0 | 0
  CREA, PII(D37), G4 | 0 | 0 | 0 | 0 | 0
  CREA, PII(D37), Missing | 2 | 3 | 52 | 2 | 2

51. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: Seven days post Dose 3 [PIII(D67)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 49 | 52 | 49
Participants
  Haem, PIII(D67), Normal | 46 | 51 | 46
  Haem, PIII(D67), G1 | 0 | 0 | 0
  Haem, PIII(D67), G2 | 0 | 0 | 0
  Haem, PIII(D67), G4 | 0 | 0 | 0
  Haem, PIII(D67), Missing | 3 | 1 | 3
  WBC, PIII(D67), Normal | 44 | 49 | 46
  WBC, PIII(D67), G1 | 0 | 0 | 0
  WBC, PIII(D67), G2 | 0 | 0 | 0
  WBC, PIII(D67), G4 | 0 | 0 | 0
  WBC, PIII(D67), Missing | 5 | 3 | 3
  PLA, PIII(D67), Normal | 46 | 51 | 46
  PLA, PIII(D67), G1 | 0 | 0 | 0
  PLA, PIII(D67), G2 | 0 | 0 | 0
  PLA, PIII(D67), G4 | 0 | 0 | 0
  PLA, PIII(D67), Missing | 3 | 1 | 3
  ALA, PIII(D67), Normal | 46 | 51 | 45
  ALA, PIII(D67), G1 | 0 | 1 | 0
  ALA, PIII(D67), G2 | 0 | 0 | 0
  ALA, PIII(D67), G4 | 0 | 0 | 0
  ALA, PIII(D67), Missing | 3 | 0 | 4
  CREA, PIII(D67), Normal | 46 | 52 | 45
  CREA, PIII(D67), G1 | 0 | 0 | 0
  CREA, PIII(D67), G2 | 0 | 0 | 0
  CREA, PIII(D67), G4 | 0 | 0 | 0
  CREA, PIII(D67), Missing | 3 | 0 | 4

52. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: One Month post Dose 1 [PI(M1)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50 | 50
Participants
  Haem, PI(M1), Normal | 0 | 45 | 0
  Haem, PI(M1), G1 | 0 | 2 | 0
  Haem, PI(M1), G2 | 0 | 0 | 0
  Haem, PI(M1), G4 | 0 | 0 | 0
  Haem, PI(M1), Missing | 50 | 3 | 50
  WBC, PI(M1), Normal | 0 | 46 | 0
  WBC, PI(M1), G1 | 0 | 0 | 0
  WBC, PI(M1), G2 | 0 | 0 | 0
  WBC, PI(M1), G4 | 0 | 0 | 0
  WBC, PI(M1), Missing | 50 | 4 | 50
  PLA, PI(M1), Normal | 0 | 47 | 0
  PLA, PI(M1), G1 | 0 | 0 | 0
  PLA, PI(M1), G2 | 0 | 0 | 0
  PLA, PI(M1), G4 | 0 | 0 | 0
  PLA, PI(M1), Missing | 50 | 3 | 50
  ALA, PI(M1), Normal | 0 | 42 | 0
  ALA, PI(M1), G1 | 0 | 0 | 0
  ALA, PI(M1), G2 | 0 | 0 | 0
  ALA, PI(M1), G4 | 0 | 0 | 0
  ALA, PI(M1), Missing | 50 | 8 | 50
  CREA, PI(M1), Normal | 0 | 42 | 0
  CREA, PI(M1), G1 | 0 | 0 | 0
  CREA, PI(M1), G2 | 0 | 0 | 0
  CREA, PI(M1), G4 | 0 | 0 | 0
  CREA, PI(M1), Missing | 50 | 8 | 50

53. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: One Month post Dose 2 [PII(M2)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50
Participants
  Haem, PII(M2), Normal | 47 | 44
  Haem, PII(M2), G1 | 0 | 0
  Haem, PII(M2), G2 | 0 | 0
  Haem, PII(M2), G4 | 0 | 0
  Haem, PII(M2), Missing | 3 | 6
  WBC, PII(M2), Normal | 45 | 41
  WBC, PII(M2), G1 | 0 | 0
  WBC, PII(M2), G2 | 0 | 0
  WBC, PII(M2), G4 | 0 | 0
  WBC, PII(M2), Missing | 5 | 9
  PLA, PII(M2), Normal | 47 | 44
  PLA, PII(M2), G1 | 0 | 0
  PLA, PII(M2), G2 | 0 | 0
  PLA, PII(M2), G4 | 0 | 0
  PLA, PII(M2), Missing | 3 | 6
  ALA, PII(M2), Normal | 42 | 36
  ALA, PII(M2), G1 | 0 | 0
  ALA, PII(M2), G2 | 0 | 0
  ALA, PII(M2), G4 | 0 | 0
  ALA, PII(M2), Missing | 8 | 14
  CREA, PII(M2), Normal | 42 | 36
  CREA, PII(M2), G1 | 0 | 0
  CREA, PII(M2), G2 | 0 | 0
  CREA, PII(M2), G4 | 0 | 0
  CREA, PII(M2), Missing | 8 | 14

54. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: One Month post Dose 3 [PIII(M3)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 49 | 52 | 49
Participants
  Haem, PIII(M3), Normal | 46 | 49 | 44
  Haem, PIII(M3), G1 | 0 | 0 | 0
  Haem, PIII(M3), G2 | 0 | 0 | 0
  Haem, PIII(M3), G4 | 0 | 0 | 0
  Haem, PIII(M3), Missing | 3 | 3 | 5
  WBC, PIII(M3), Normal | 45 | 48 | 43
  WBC, PIII(M3), G1 | 0 | 0 | 0
  WBC, PIII(M3), G2 | 0 | 0 | 0
  WBC, PIII(M3), G4 | 0 | 0 | 0
  WBC, PIII(M3), Missing | 4 | 4 | 6
  PLA, PIII(M3), Normal | 46 | 48 | 44
  PLA, PIII(M3), G1 | 0 | 0 | 0
  PLA, PIII(M3), G2 | 0 | 0 | 0
  PLA, PIII(M3), G4 | 0 | 0 | 0
  PLA, PIII(M3), Missing | 3 | 3 | 5
  ALA, PIII(M3), Normal | 46 | 50 | 44
  ALA, PIII(M3), G1 | 0 | 0 | 0
  ALA, PIII(M3), G2 | 0 | 0 | 0
  ALA, PIII(M3), G4 | 0 | 0 | 0
  ALA, PIII(M3), Missing | 3 | 2 | 5
  CREA, PIII(M3), Normal | 46 | 50 | 44
  CREA, PIII(M3), G1 | 0 | 0 | 0
  CREA, PIII(M3), G2 | 0 | 0 | 0
  CREA, PIII(M3), G4 | 0 | 0 | 0
  CREA, PIII(M3), Missing | 3 | 2 | 5

55. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 49
Time Frame: Six Months post Dose 1 [PI(M6)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 1 Dose Group
Number analyzed (Participants) | 50
Participants
  Haem, PI(M6), Normal | 41
  Haem, PI(M6), G1 | 4
  Haem, PI(M6), G2 | 1
  Haem, PI(M6), G4 | 0
  Haem, PI(M6), Missing | 4
  WBC, PI(M6), Normal | 45
  WBC, PI(M6), G1 | 0
  WBC, PI(M6), G2 | 0
  WBC, PI(M6), G4 | 0
  WBC, PI(M6), Missing | 5
  PLA, PI(M6), Normal | 46
  PLA, PI(M6), G1 | 0
  PLA, PI(M6), G2 | 0
  PLA, PI(M6), G4 | 0
  PLA, PI(M6), Missing | 4
  ALA, PI(M6), Normal | 45
  ALA, PI(M6), G1 | 1
  ALA, PI(M6), G2 | 0
  ALA, PI(M6), G4 | 0
  ALA, PI(M6), Missing | 4
  CREA, PI(M6), Normal | 46
  CREA, PI(M6), G1 | 0
  CREA, PI(M6), G2 | 0
  CREA, PI(M6), G4 | 0
  CREA, PI(M6), Missing | 4

56. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: Six Months post Dose 2 [PII(M7)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50
Participants
  Haem, PII(M7), Normal | 42 | 41
  Haem, PII(M7), G1 | 3 | 3
  Haem, PII(M7), G2 | 0 | 0
  Haem, PII(M7), G4 | 0 | 0
  Haem, PII(M7), Missing | 5 | 6
  WBC, PII(M7), Normal | 42 | 44
  WBC, PII(M7), G1 | 0 | 0
  WBC, PII(M7), G2 | 0 | 0
  WBC, PII(M7), G4 | 0 | 0
  WBC, PII(M7), Missing | 8 | 6
  PLA, PII(M7), Normal | 45 | 44
  PLA, PII(M7), G1 | 0 | 0
  PLA, PII(M7), G2 | 0 | 0
  PLA, PII(M7), G4 | 0 | 0
  PLA, PII(M7), Missing | 5 | 6
  ALA, PII(M7), Normal | 43 | 43
  ALA, PII(M7), G1 | 0 | 0
  ALA, PII(M7), G2 | 0 | 0
  ALA, PII(M7), G4 | 0 | 0
  ALA, PII(M7), Missing | 7 | 7
  CREA, PII(M7), Normal | 43 | 43
  CREA, PII(M7), G1 | 0 | 0
  CREA, PII(M7), G2 | 0 | 0
  CREA, PII(M7), G4 | 0 | 0
  CREA, PII(M7), Missing | 7 | 7

57. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: Six Months post Dose 3 [PIII(M8)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 49 | 52 | 49
Participants
  Haem, PIII(M8), Normal | 43 | 47 | 44
  Haem, PIII(M8), G1 | 1 | 4 | 2
  Haem, PIII(M8), G2 | 0 | 0 | 0
  Haem, PIII(M8), G4 | 0 | 0 | 0
  Haem, PIII(M8), Missing | 5 | 1 | 3
  WBC, PIII(M8), Normal | 41 | 47 | 41
  WBC, PIII(M8), G1 | 0 | 0 | 0
  WBC, PIII(M8), G2 | 0 | 0 | 0
  WBC, PIII(M8), G4 | 0 | 0 | 0
  WBC, PIII(M8), Missing | 8 | 5 | 8
  PLA, PIII(M8), Normal | 44 | 50 | 46
  PLA, PIII(M8), G1 | 0 | 1 | 0
  PLA, PIII(M8), G2 | 0 | 0 | 0
  PLA, PIII(M8), G4 | 0 | 0 | 0
  PLA, PIII(M8), Missing | 5 | 1 | 3
  ALA, PIII(M8), Normal | 43 | 50 | 46
  ALA, PIII(M8), G1 | 1 | 0 | 0
  ALA, PIII(M8), G2 | 0 | 0 | 0
  ALA, PIII(M8), G4 | 0 | 0 | 0
  ALA, PIII(M8), Missing | 5 | 1 | 3
  CREA, PIII(M8), Normal | 43 | 51 | 46
  CREA, PIII(M8), G1 | 0 | 0 | 0
  CREA, PIII(M8), G2 | 0 | 0 | 0
  CREA, PIII(M8), G4 | 0 | 0 | 0
  CREA, PIII(M8), Missing | 6 | 1 | 3

58. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: Six Months post Dose 3 [PIII(M13)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50
Participants
  Haem, PIII(M13), Normal | 0 | 43
  Haem, PIII(M13), G1 | 0 | 1
  Haem, PIII(M13), G2 | 0 | 0
  Haem, PIII(M13), G4 | 0 | 0
  Haem, PIII(M13), Missing | 50 | 6
  WBC, PIII(M13), Normal | 0 | 42
  WBC, PIII(M13), G1 | 0 | 0
  WBC, PIII(M13), G2 | 0 | 0
  WBC, PIII(M13), G4 | 0 | 0
  WBC, PIII(M13), Missing | 50 | 8
  PLA, PIII(M13), Normal | 0 | 44
  PLA, PIII(M13), G1 | 0 | 0
  PLA, PIII(M13), G2 | 0 | 0
  PLA, PIII(M13), G4 | 0 | 0
  PLA, PIII(M13), Missing | 50 | 6
  ALA, PIII(M13), Normal | 0 | 44
  ALA, PIII(M13), G1 | 0 | 0
  ALA, PIII(M13), G2 | 0 | 0
  ALA, PIII(M13), G4 | 0 | 0
  ALA, PIII(M13), Missing | 50 | 6
  CREA, PIII(M13), Normal | 0 | 44
  CREA, PIII(M13), G1 | 0 | 0
  CREA, PIII(M13), G2 | 0 | 0
  CREA, PIII(M13), G4 | 0 | 0
  CREA, PIII(M13), Missing | 50 | 6

59. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: Twelve Months post Dose 1 [PI(M12)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 1 Dose Group
Number analyzed (Participants) | 50
Participants
  Haem, PI(M12), Normal | 47
  Haem, PI(M12), G1 | 2
  Haem, PI(M12), G2 | 0
  Haem, PI(M12), G4 | 0
  Haem, PI(M12), Missing | 1
  WBC, PI(M12), Normal | 48
  WBC, PI(M12), G1 | 0
  WBC, PI(M12), G2 | 0
  WBC, PI(M12), G4 | 0
  WBC, PI(M12), Missing | 2
  PLA, PI(M12), Normal | 48
  PLA, PI(M12), G1 | 1
  PLA, PI(M12), G2 | 0
  PLA, PI(M12), G4 | 0
  PLA, PI(M12), Missing | 1
  ALA, PI(M12), Normal | 46
  ALA, PI(M12), G1 | 2
  ALA, PI(M12), G2 | 1
  ALA, PI(M12), G4 | 0
  ALA, PI(M12), Missing | 1
  CREA, PI(M12), Normal | 49
  CREA, PI(M12), G1 | 0
  CREA, PI(M12), G2 | 0
  CREA, PI(M12), G4 | 0
  CREA, PI(M12), Missing | 1

60. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: Twelve Months post Dose 2 [PII(M13)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692342 2 Dose Group | Control Menjugate Group
Number analyzed (Participants) | 50 | 50
Participants
  Haem, PII(M13), Normal | 41 | 0
  Haem, PII(M13), G1 | 4 | 0
  Haem, PII(M13), G2 | 1 | 0
  Haem, PII(M13), G4 | 0 | 0
  Haem, PII(M13), Missing | 4 | 50
  WBC, PII(M13), Normal | 43 | 0
  WBC, PII(M13), G1 | 0 | 0
  WBC, PII(M13), G2 | 0 | 0
  WBC, PII(M13), G4 | 0 | 0
  WBC, PII(M13), Missing | 7 | 50
  PLA, PII(M13), Normal | 46 | 0
  PLA, PII(M13), G1 | 0 | 0
  PLA, PII(M13), G2 | 0 | 0
  PLA, PII(M13), G4 | 0 | 0
  PLA, PII(M13), Missing | 4 | 50
  ALA, PII(M13), Normal | 45 | 0
  ALA, PII(M13), G1 | 1 | 0
  ALA, PII(M13), G2 | 0 | 0
  ALA, PII(M13), G4 | 0 | 0
  ALA, PII(M13), Missing | 4 | 50
  CREA, PII(M13), Normal | 46 | 0
  CREA, PII(M13), G1 | 0 | 0
  CREA, PII(M13), G2 | 0 | 0
  CREA, PII(M13), G4 | 0 | 0
  CREA, PII(M13), Missing | 4 | 50

61. Secondary Outcome: Number of Subjects With Normal, G1, G2, or G4 Haematological and Biochemical Markers
Description: as for outcome 50
Time Frame: Twelve Months post Dose 3 [PIII(M14)]
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
Number analyzed (Participants) | 49 | 52 | 49
Participants
  Haem, PIII(M14), Normal | 38 | 46 | 37
  Haem, PIII(M14), G1 | 6 | 5 | 8
  Haem, PIII(M14), G2 | 0 | 0 | 0
  Haem, PIII(M14), G4 | 0 | 0 | 0
  Haem, PIII(M14), Missing | 5 | 1 | 4
  WBC, PIII(M14), Normal | 42 | 48 | 42
  WBC, PIII(M14), G1 | 0 | 0 | 0
  WBC, PIII(M14), G2 | 0 | 0 | 0
  WBC, PIII(M14), G4 | 0 | 0 | 0
  WBC, PIII(M14), Missing | 7 | 4 | 7
  PLA, PIII(M14), Normal | 44 | 51 | 44
  PLA, PIII(M14), G1 | 0 | 0 | 0
  PLA, PIII(M14), G2 | 0 | 0 | 0
  PLA, PIII(M14), G4 | 0 | 0 | 0
  PLA, PIII(M14), Missing | 5 | 1 | 4
  ALA, PIII(M14), Normal | 43 | 51 | 43
  ALA, PIII(M14), G1 | 1 | 0 | 1
  ALA, PIII(M14), G2 | 0 | 0 | 0
  ALA, PIII(M14), G4 | 0 | 0 | 0
  ALA, PIII(M14), Missing | 5 | 1 | 5
  CREA, PIII(M14), Normal | 44 | 51 | 44
  CREA, PIII(M14), G1 | 0 | 0 | 0
  CREA, PIII(M14), G2 | 0 | 0 | 0
  CREA, PIII(M14), G4 | 0 | 0 | 0
  CREA, PIII(M14), Missing | 5 | 1 | 5

ADVERSE EVENTS:
Time Frame: Solicited symptoms: during the 7-day post-vaccination period; Unsolicited AEs: during the 30-day post-vaccination period; SAEs: from study start (Day 0) up to one month post-vaccination and from Day 0 up to 12 months post last vaccination.
Description: Other Adverse Events were collected from all subjects with at least one administered dose with safety follow-up and who completed their symptom sheet.
Arm/Group | SB692342 2 Dose Group | SB692342 1 Dose Group | Control Menjugate Group | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group | Control Tritanrix + Prevnar + Polio Sabin Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 1/50 | 0/49 | 0/52 | 0/49
Serious Adverse Events (participants affected / at risk) | 2/50 | 3/50 | 3/50 | 1/49 | 1/52 | 1/49
Other Adverse Events (participants affected / at risk) | 33/50 | 22/50 | 31/50 | 34/49 | 22/52 | 26/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB692342 2 Dose Group (N=50) | SB692342 1 Dose Group (N=50) | Control Menjugate Group (N=50) | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group (N=49) | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group (N=52) | Control Tritanrix + Prevnar + Polio Sabin Group (N=49)
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0
Cerebral malaria (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Malaria (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SB692342 2 Dose Group (N=50) | SB692342 1 Dose Group (N=50) | Control Menjugate Group (N=50) | SB692392 2 Dose + Tritanrix + Prevnar + Polio Sabin Group (N=49) | SB692392 1 Dose + Tritanrix + Prevnar + Polio Sabin Group (N=52) | Control Tritanrix + Prevnar + Polio Sabin Group (N=49)
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 3
Pyrexia (General disorders) | 3 | 1 | 4 | 0 | 2 | 0
Pain (General disorders) | 6 | 2 | 6 | 10 | 13 | 13
Swelling (General disorders) | 0 | 0 | 0 | 6 | 8 | 8
Drowsiness (General disorders) | 2 | 0 | 1 | 3 | 3 | 0
Irritability (General disorders) | 3 | 0 | 2 | 8 | 5 | 4
Loss of appetite (General disorders) | 3 | 0 | 1 | 3 | 2 | 0
Temperature (Axillary) (General disorders) | 19 | 5 | 13 | 18 | 9 | 12
Diarrhoea (Gastrointestinal disorders) | 8 | 5 | 2 | 5 | 1 | 3
Respiratory tract infection (Infections and infestations) | 21 | 14 | 19 | 15 | 9 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.